CLINICAL TRIAL: NCT06806865
Title: Comparison of Continuous Fascia Iliaca Compartment Block With Continuous PENG Block in Total Hip Replacement Cases
Acronym: PENG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Ayhan ŞAHİN, Assistant Professor, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023.06.01.06
Record Dates: First submitted 2024-12-30; First posted 2025-02-04 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain; Regional Anesthesia; Pain Management; Total Hip Arthroplasty
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants will be randomly divided into two groups. The physician who will collect data in the orthopedic department will not know which group the participant is in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENG Group (periarticular nerve group) (Active Comparator): Continuous PENG block is the group to be applied.
  Interventions: Procedure: Periarticular nerve group block (PENG)
- SIFICB Group (supra-inguinal fascia iliaca compartment block) (Active Comparator): Continuous supra-inguinal fascia iliaca compartment block is the group to be applied.
  Interventions: Procedure: Continuous supra-inguinal fascia iliaca compartment block (SIFICB)

INTERVENTIONS:
Procedure: Periarticular nerve group block (PENG) — The pericapsular nerve group (PENG) block targets the nerves that supply the hip capsule. The continuous PENG block will be applied immediately after general anesthesia is given to the participants under ultrasound guidance. 30 ml of 0.25% bupivacaine will be used.
  Arms: PENG Group (periarticular nerve group)
Procedure: Continuous supra-inguinal fascia iliaca compartment block (SIFICB) — The supra-inguinal fascia iliaca compartment block (SIFICB) targets the femoral, lateral femoral cutaneous, and obturator nerves. Under ultrasound guidance, 30 mL of 0.25% bupivacaine is administered, followed by catheter placement for continuous infusion at 5 mL/h.
  Arms: SIFICB Group (supra-inguinal fascia iliaca compartment block)

SUMMARY:
Adequate pain management after total hip arthroplasty (THA) is crucial for early ambulation and patient satisfaction. However, due to the hip joint's innervation complexity, the optimal regional analgesia technique for THA remains controversial.

Total hip arthroplasties are critical surgeries that can take steps to improve the quality of life and functional status of patients who do not respond to conservative treatments. However, patients may present with intense pain in the immediate postoperative period, resulting in inactivity, increased risk of complications, and greater opioid consumption, resulting in adverse effects and prolonged hospital stay. The challenging management of pain is explained by the complex innervation of the hip joint, in which the articular branches of the femoral, obturator, and accessory obturator nerves are responsible for the sensory innervation of the anterior capsule.

This randomized clinical trial compares the analgesic efficacy of FICB and PENG block following THA. Our preliminary results will be postoperative pain scores. As our anesthesia clinic, we routinely perform these known methods after surgery in these cases. Traditional intravenous analgesia methods cause many undesirable side effects depending on the type of opioid used, and they are insufficient compared to regional anesthesia methods.

DETAILED DESCRIPTION:
The pericapsular nerve group (PENG) block has been reported as the first method to target the nerves that supply the hip capsule. Later, several studies said it was more effective than traditional peripheral nerve blocks at treating THA-related postoperative pain. However, a single-injection PENG block is only effective for a limited time. Little evidence supports the efficacy of continuous PENG block for postoperative pain management in THA.

Additional anesthetic techniques, such as peripheral nerve blocks, are part of the multimodal analgesic strategy and are often used to manage acute pain better. Inadequate treatment can lead to a persistent painful condition. Although numerous nerve blocks are available for this purpose, some may fail because they cover only some of the innervation of the anterior hip capsule. The trial hypothesizes that with continuous infusion of the pericapsular nerve group block (PENG block), defined in 2018, the four lateral cutaneous nerve blocks local anesthetic between the thigh-associated psoas muscle tendon plane, and the iliopubic eminence will provide adequate analgesia without causing a motor block. Compared to the infrainguinal approach, the fascia iliaca compartment block (FICB) provides better dissemination under the fascia iliaca, while the local anesthetic is administered more cranially. Desmet et al. showed that supra-inguinal FICB reduced morphine consumption and pain scores following THA. However, despite these promising results, obturator nerve block has not been clinically proven.

Total hip arthroplasties are necessary surgeries that can take steps to improve the quality of life and functional status of patients who do not respond to conservative treatments. However, patients may present with intense pain in the immediate postoperative period, resulting in inactivity, increased risk of complications, and greater opioid consumption, resulting in adverse effects and prolonged hospital stay. The challenging management of pain is explained by the complex innervation of the hip joint, in which the articular branches of the femoral, obturator, and accessory obturator nerves are responsible for the sensory innervation of the anterior capsule.

This randomized clinical trial hypothesizes that PENG block will provide better analgesia and result in fewer quadriceps muscle weakness than FICB following THA. Our preliminary results will be postoperative pain scores. Most anesthesia clinics routinely do this by diversifying these methods known after surgery. Traditional intravenous analgesia methods cause many undesirable side effects depending on the type of opioid used, and they are insufficient compared to regional anesthesia methods.

Since THA patients are generally elderly and with comorbidities, regional anesthesia techniques are safer and more effective.

This study focuses on two routine regional anesthesia techniques that can be safely applied. The trial aims to show which of these two methods is more effective.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing hip replacement for the first time
2. Patients aged 18-65 years, ASAI-II (American Society of Anesthesiology classification)
3. Patients without primary cancer and/or patients without metastatic bone fractures
4. Patients without allergy to local anaesthetics
5. Patients with an intellectual level that can use patient-controlled analgesia devices
6. Patients with a standard bleeding profile
7. Patients who gave written consent to participate in the study

Exclusion Criteria:

1. patients who have had a hip replacement and/or revision
2. patients who have primary cancer and/or fractures due to bone metastasis
3. patients who have a local anaesthetic allergy and/or a history of it
4. patients who are not intellectually competent enough to use a patient-controlled anesthesia device
5. patients who have undergone reoperation due to any surgical complication (bleeding, etc.) within 24 hours after surgery
6. patients who did not give written consent to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
VAS scores | up to 24 hours after recovery unit
  The Visual Analogue Scale (VAS) measures pain intensity. It consists of a 10 cm line with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could be'). Ask the patient to rate their current level of pain by placing a mark on the line. VAS scores at rest and during movement will be recorded at 0 hours (PACU), and subsequently at 2, 6, 12, and 24 hours while the patient is in the orthopedic clinic.

SECONDARY OUTCOMES:
Total patient-controlled analgesia (PCA) consumption for 24 hours postoperatively | Up to 24 hours
  A patient-controlled analgesia (PCA) pump is a safe way for people in pain to administer intravenous (I.V.) pain medicine (analgesia) when they need it. The pump holds a container filled with pain medicine, allowing the patient to control their pain. A total of 300 mg of tramadol will be used. 3mg/cc.
intraoperative blood pressure | from the beginning of anesthesia induction to the leaving the recovery unit
  Blood pressure will be monitored and recorded intermittently throughout the surgery. These parameters may be signs of pain.
need for additional analgesia or rescue analgesia | up to 24 hours after surgery
  In cases where pain control is inadequate, when the PCA is locked and the VAS score is five or above, additional analgesics are administered. Paracetamol 15 mg/kg will be administered as rescue analgesia in the study.
intraoperative heart rate | from the beginning of anesthesia induction up to leaving the recovery unit
  Heart rate will be monitored and recorded intermittently throughout the surgery. These parameters may be signs of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Namık Kemal Üniversitesi, Tekirdağ, Süleymanpasa, Turkey (Türkiye)

REFERENCES:
- [Derived] Baran O, Sahin A, Arar C. Comparative analysis of continuous pericapsular nerve group block and supra-inguinal fascia iliaca compartment block for postoperative analgesia in total hip arthroplasty: a randomized controlled trial. J Orthop Surg Res. 2025 Aug 6;20(1):729. doi: 10.1186/s13018-025-06055-w. PMID 40770360